CLINICAL TRIAL: NCT02991157
Title: Noninvasive Assessment of Cerebral Oxygenation and Cardiac Function in Patients With Neurovascular Diseases
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Sriganesh Kamath, Associate Professor, National Institute of Mental Health and Neuro Sciences, India
Other Study IDs: 12.02
Record Dates: First submitted 2016-12-07; First posted 2016-12-13 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: cerebral vasospasm; nimodipine
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — Nimodipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Nimodipine

SUMMARY:
This prospective observational study will assess the regional cerebral oxygen saturation and cardiac output non-invasively in patients with subarachnoid hemorrhage during nimodipine administration for the prevention/management of cerebral vasospasm.

ELIGIBILITY:
Inclusion Criteria:

* aneurysmal subarachnoid hemorrhage
* potential or actual cerebral vasospasm

Exclusion Criteria:

* non-aneurysmal subarachnoid hemorrhage
* outside the 4-21 day window after ictus
* peripheral deoxygenation
* contraindication for nimodipine administration

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: aneurysmal subarachnoid hemorrhage with cerebral vasospasm
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in the cerebral oxygen saturation percentage measured using near infrared spectroscopy technology after administration of nimodipine | Change from baseline cerebral oxygen saturation at 30 minutes after administration of nimodipine

SECONDARY OUTCOMES:
Change in the cardiac output measured using near NICOM technology after administration of nimodipine | Change from baseline cardiac output at 30 and 240 minutes after administration of nimodipine
  unit of measurement will be L/min
Change in the cerebral oxygen saturation percentage measured using near infrared spectroscopy technology after administration of nimodipine | Change from baseline cerebral oxygen saturation at 240 minutes after administration of nimodipine

CONTACTS AND LOCATIONS:
Locations (1):
- NIMHANS, Bengaluru, India